CLINICAL TRIAL: NCT02647437
Title: Effects of Low-dose Levetiracetam on Clinical Symptoms, Cognition and Hippocampal Hyperactivity in Patients With Schizophrenia
Brief Title: Effects of Low-dose Levetiracetam on Clinical Symptoms, Cognition and Hippocampal Hyperactivity in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 13-1495
Record Dates: First submitted 2015-12-29; First posted 2016-01-06 (Estimated); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Levetiracetam

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levetiracetam, Then Placebo (Experimental): 2 weeks of levetiracetam administration (125 mg pill, bid), followed by a 1-2 week washout, then 2 weeks of placebo pill administration (bid).
  Interventions: Drug: Levetiracetam; Drug: Placebo
- Placebo, Then Levetiracetam (Experimental): 2 weeks of placebo pill administration (bid), followed by a 1-2 week washout, then 2 weeks of levetiracetam administration (125 mg pill, bid).
  Interventions: Drug: Levetiracetam; Drug: Placebo

INTERVENTIONS:
Drug: Levetiracetam
  Other Names: Keppra
Drug: Placebo

SUMMARY:
Levetiracetam (LEV: (S)-α-ethyl-2-oxo-pyrrolidine acetamide) is an anticonvulsant/antiepileptic drug. The specific aim of this study is to assess the efficacy of low-dose LEV in reducing hippocampal activity in schizophrenia. The investigators also hypothesize that LEV will improve neurocognition in participants with schizophrenia.

DETAILED DESCRIPTION:
LEV is typically administered in twice-daily doses of 500-1500 mg for the treatment of epilepsy; these doses are generally well tolerated (Patsalos, 2000). Most relevant to the proposed study, LEV (125 mg twice-daily, two week administration) has been shown to reduce hippocampal hyperactivity and improves cognition in patients with mild cognitive impairment (MCI).

The proposed study will administer 125 mg of immediate release LEV twice-daily for two weeks. This dose was chosen to potentially maximize efficacy while minimizing side effects. The proposed dose is substantially lower than the most common dose used clinically for epilepsy treatment of 3000 mg/day.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizoaffective disorder
* Good general health
* Normal vital signs (blood pressure, pulse, cardiac, pulmonary, abdominal, neurological exam)
* Normal renal function (as assessed by a metabolic panel at screening if results current within three months are not already available)

Exclusion Criteria:

1. Substance abuse
2. Significant neurological disorders
3. Significant head trauma/injury
4. Left-handedness
5. Pregnancy
6. MRI-specific exclusion criteria (e.g., claustrophobia, weight > 450lbs, metal in the body)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-06; Primary Completion 2024-09 (Actual); Study Completion 2024-09 (Actual)

PRIMARY OUTCOMES:
Resting-state neuronal response | 2 weeks
  Neuronal response (measured via functional magnetic resonance imaging, fMRI) in the hippocampus during rest

SECONDARY OUTCOMES:
Neurocognitive function | 2 weeks
  Cognitive function as measured by the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Tregellas, Ph.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No